CLINICAL TRIAL: NCT02179554
Title: Does Cardiopulmonary Bypass Change Olfaction?
Acronym: Anosmia
Status: Withdrawn | Type: Observational
Sponsor: Manchester University NHS Foundation Trust (Other Government)
Responsible Party: Sponsor
Other Study IDs: R03463
Record Dates: First submitted 2014-06-25; First posted 2014-07-02 (Estimated); Last update posted 2020-03-17 (Actual); Status verified 2020-03

CONDITIONS: Anosmia
MeSH Terms: conditions — Anosmia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- cardiopulmonary bypass: Patients undergoing elective surgery requiring cardiopulmonary bypass

SUMMARY:
The loss of the sense of smell, anosmia, can have profound effects on the lives of those who suffer from it. In our clinical practice, we have encountered several patients complaining of anosmia after recently undergoing surgery requiring cardiopulmonary bypass. We want to investigate this peculiar observation and determine if such a link exists. Thus far, there have been no similar studies published, and as such, no previous evidence on this matter. This study will help formalise and clarify these observations, empowering clinicians to better inform patients in the future; if cardiopulmonary bypass procedures do carry a risk of anosmia. This study may also give rise to further research into the matter.

DETAILED DESCRIPTION:
Objectives: To investigate the incidence of anosmia arising in patients after undergoing cardiopulmonary bypass, and compare it to a control group.

Hypothesis: Patients undergoing cardiopulmonary bypass may suffer from anosmia.

Methodology: Potential participants will be identified via scheduled operating lists at Manchester Royal Infirmary. Suitable patients will be informed, including informational leaflets about the study, and permissions sought with an informed consent form. Once recruited, when the patients come for their pre-operative assessment, olfactory assessment will be carried out using the Sniffing Sticks smell kit and a validated questionnaire (Dresden Questionnaire of Olfactory Disorders). The Sniffing Sticks smell kit composes of 12 different pen-like odour dispensers. Each stick is presented to the patient who then chooses from four different answers, the one that best represents the odour. The patient then receives a score of 0 to 12. A reassessment via the same questionnaire and smell kit is repeated after 1 week or just before discharge (whichever is earlier) after the patient's surgery.

Data Management and Statistical Analyses: All participant information will be stored electronically in a password protected trust computer. Participant identifiers will also be kept in a separate password protected folder from the main database of individual participant information. We will use MS Excel for compiling the data.

Study Type: Prospective, single-centre, observational study

Target Sample size: 50 patients undergoing elective surgery requiring cardiopulmonary bypass (study group) 50 patients total

Procedures for Obtaining and Documenting Consent: All patients undergoing major surgery will require to attend a preoperative planning clinic. Information leaflets will be disseminated at this time, which includes contact details of involved researchers. Depending on availability, the principal researcher would be present during the preoperative clinics to answer any questions. Contact details will be taken for any patient considering to participate at this point whilst any patient who initially refuse and choose to participate later will require to contact the researchers to opt back in. Potential participants will then be contacted via their mode of choice (email/telephone) to assess if they want to participate. On the day of planned admission into hospital for elective surgery, or at another agreed upon time, a written consent will be obtained and all questions addressed immediately before the study is conducted. Patients undergoing major surgery are normally admitted into hospital the day before surgery. This time period is opportunistic as from experience, most patients will have ample free time from then till the day of surgery and a distraction would most probably be welcome. However, if no such opportunity is foreseen, a separate appointment in hospital grounds can be made at a suitable time. After the operation, a repeat study will be done, ideally in conjunction with any one of their follow up visits to the hospital, which normally involves a waiting time. Otherwise, an alternate suitable appointment can be arranged. Any arranged appointments will restricted to working hours (Mon-Fri 8am-5pm) in the ENT outpatients department at Manchester Royal Infirmary.

Risks and benefits: There are no risks to patients who participate in this study. There are also no direct benefits to the participant other than having a free objective measurement of their sense of smell and learning about the nature of the study. Patient participation is purely voluntary.

Confidentiality: Each participant will be identified by an assigned code number. This will be stored in a separate file from the main database, only accessible on a password protected server. Thus, each participant's data is kept anonymous. Informed consent forms will be locked a separate file cabinet.

ELIGIBILITY:
Inclusion Criteria:

- English speaking volunteers above 18 years of age.

Exclusion Criteria:

- Pre-existing olfaction disorder, nasal polyps.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 50 patients undergoing elective surgery requiring cardiopulmonary bypass (study group)
Sampling Method: Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2014-10; Primary Completion 2015-10 (Estimated); Study Completion 2015-12 (Estimated)

PRIMARY OUTCOMES:
1) Sniffin sticks score out of 16 | 1 day
  1) Objective scoring based smell test kit

SECONDARY OUTCOMES:
2) Dresden questionnaire of olfactory disorder score | 1 day
  2) Scoring based on validated questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Atef El-Kholy, Principal Investigator — Manchester University NHS Foundation Trust
Locations (1):
- Central Manchester University Hospitals NHS Foundation Trust, Manchester, Greater Manchester, United Kingdom